CLINICAL TRIAL: NCT00202969
Title: An Open-label, Multicenter, Randomized, 3 Arm Study of S-1 Compared With S-1/CDDP, or S-1/CDDP Compared With 5-FU/CDDP in Patients With Advanced Gastric Cancer Previously Untreated With Chemotherapy for Advanced Disease
Brief Title: Study of S-1, S-1/CDDP, and 5-FU/CDDP for Advanced Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Taiho Pharmaceutical Co., Ltd., Taiho Pharmaceutical Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SC101
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Gastric Cancer
Keywords: Stomach cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); Fluorouracil

ARMS (3):
- 1 (Experimental): S-1
  Interventions: Drug: S-1
- 2 (Active Comparator): S-1 plus CDDP
  Interventions: Drug: S-1 plus CDDP
- 3 (Active Comparator): 5-FU plus CDDP
  Interventions: Drug: 5-FU plus CDDP

INTERVENTIONS:
Drug: S-1 — S-1 40 mg/m2 administered orally BID after breakfast and evening meal from Day 1 through Day 28 repeated 6 weeks.
  Arms: 1
Drug: S-1 plus CDDP — S-1 40 mg/m2 administered orally BID after breakfast and evening meal from Day 1 through Day 21 with a single dose of CDDP 60 mg/m2 will be administered as an 1- to 3-hour IV infusion following the morning dose of S-1 on Day 8. The combination therapy will be repeated every 5 weeks.
  Arms: 2
Drug: 5-FU plus CDDP — 5-FU 600 mg/m2/24 hours administered intravenously as a CI over 120 hours (Days 1 through 5) along with a 30-minute infusion CDDP 20 mg/m2 from Day 1 through Day 5. The control treatment arm will be repeated every 4 weeks.
  Arms: 3

SUMMARY:
This is an open-label, multicenter, three arm, parallel, randomized, Phase 3 study evaluating the efficacy and safety of S-1 alone compared with S-1 plus CDDP, and S-1 plus CDDP compared with 5-FU plus CDDP in patients with advanced gastric cancer previously untreated with chemotherapy for advanced disease. Patients will be randomly assigned (1:1:1) to S-1 (Arm A), S-1/CDDP (Arm B) or 5-FU/CDDP (Arm C). Patients will be stratified to achieve balanced distribution of patients to each arm according to following stratifications, performance status (0, 1, or 2), the number of metastatic sites (1 vs >1), prior gastrectomy, and center.

ELIGIBILITY:
Inclusion Criteria:

* Non-prior chemotherapy treated advanced gastric adenocarcinoma
* Age 18 and over
* Performance status 0, 1, or 2 (ECOG)
* Life expectancy 3 months
* Hematopoietic WBC lower limit of normal-12,000/mm^3 Absolute granulocyte count ≥ 2,000/mm^3 Platelet count ≥ 100,000/mm^3 Hemoglobin ≥ 8.0 g/dL
* Hepatic AST and ALT ≤ 100 U/L ALP ≤ 2 times upper limit of normal (ULN) Bilirubin ≤ 1.5 mg/dL
* Renal Plasma creatinine ≤ ULN Creatinine clearance ≥ 60 mL/min

Exclusion Criteria:

* Interstitial pneumonia, pulmonary fibrosis
* Myocardial infarction within the last 6 months, severe/unstable angina, congestive heart failure
* Intestinal paralysis, intestinal obstruction, uncontrollable diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2005-07; Primary Completion 2007-01 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Response rate | every course for first three courses, then every other course

SECONDARY OUTCOMES:
Safety profile, time to treatment failure | any time

CONTACTS AND LOCATIONS:
Overall Officials: Jin Maolin, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, No.52 Fu-Cheng Road, Hai-dian District, Beijing Municipality, China